CLINICAL TRIAL: NCT01347476
Title: Patients Aged More Than 70 Had More Aggressive Prostate Cancers and Higher Risk of Biochemical Recurrence in Korea
Brief Title: Aggressive Prostate Cancers in Elderly Patients
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Seoul National University Boramae Hospital, Seoul National University Boramae Hospital
Other Study IDs: old age prostate; elderly pts with high risk CaP
Record Dates: First submitted 2011-04-29; First posted 2011-05-04 (Estimated); Last update posted 2011-05-19 (Estimated); Status verified 2011-05

CONDITIONS: Prostatic Neoplasms
Keywords: prostate-specific antigen; radical prostatectomy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- patients older than 70 years
- patients 70 years or younger

SUMMARY:
Patients aged 70 years or older had a higher possibility of high risk cancer than younger patients.

DETAILED DESCRIPTION:
Patients aged 70 years or older had a higher risk of advanced prostate cancer and shorter BCR-free survival than younger ones. Definite treatment of clinically localized prostate cancer should be actively considered in well-selected healthy patients older than 70 years.

ELIGIBILITY:
Inclusion Criteria:

* clinically localized prostate cancer
* good health status
* follow-up period more than 12 months

Exclusion Criteria:

* insufficient clinical data
* poor health status
* clinically advanced prostate cancer

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men who underwent radical prostatectomy for the treatment of clinically localized prostate cancer
Sampling Method: Non-Probability Sample
Enrollment: 1333 (Actual)
Dates: Start 2010-01; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
biochemical recurrences (BCR) | 5 year-BCR
  BCR was defined as two consecutive increasing PSA values of more than 0.2 ng/mL

SECONDARY OUTCOMES:
pathologic outcomes | postoperative 1 week
  biopsy or pathologic Gleason scores, mean percent of positive cores and tumor volume percent, Extracapsular extension and seminal vesicle invasion

CONTACTS AND LOCATIONS:
Overall Officials: Sung Yong Cho, M.D., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Boramae Hospital, Seoul, Seoul, South Korea

REFERENCES:
- [Derived] Kim JK, Cho SY, Jeong CW, Lee SB, Ku JH, Hong SK, Byun SS, Kwak C, Him HH, Lee SE, Jeong H. Patients aged more than 70 had higher risk of locally advanced prostate cancers and biochemical recurrence in Korea. BJU Int. 2012 Aug;110(4):505-9. doi: 10.1111/j.1464-410X.2011.10927.x. Epub 2012 Feb 7. PMID 22314007